CLINICAL TRIAL: NCT00606567
Title: A Randomized Trial of Remote Monitoring of Implantable Cardioverter Defibrillators Versus Quarterly Device Interrogations in Clinic
Acronym: Medusa SAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010068; 8774 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2012-12

CONDITIONS: Tachycardia, Ventricular; Ventricular Fibrillation
Keywords: Defibrillators, Implantable
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-treatment (Active Comparator): remote monitoring with carelink every 3 months
  Interventions: Other: Methods for monitoring patients with ICD's
- 2- control (No Intervention): device interrogations in clinic every 3 months

INTERVENTIONS:
Other: Methods for monitoring patients with ICD's — Intervention comparing 2 different methods of monitoring patients with ICDs; at home monitoring vs. quarterly monitoring in the clinic.
  Arms: 1-treatment

SUMMARY:
The purpose of this study is to determine if remote monitoring of implantable cardioverter defibrillators (ICD), compared with quarterly device interrogations in clinic, will improve patients' outcomes and satisfaction and will reduce health care costs.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD), usually due to a ventricular tachyarrhythmia, is the most common cause of death in the United States. The implantable cardioverter defibrillator (ICD) has been shown to improve the survival of patients with a history of a heart attack and a weak heart (functioning at 30% or less) and those with symptomatic congestive heart failure symptoms (hearts functioning at 35% or less). Thus, the number of patients who will require ICD therapy is expected to rise exponentially over the next several years. To facilitate the follow-up of patients with ICDs, device companies have launched systems for remote monitoring of these devices. One such system is the Medtronic Carelink Monitor. Although this system has been proven in a multicenter, prospective study to be easy to use, it is not known whether this monitor results in improved patients' outcomes and satisfaction and in reduced healthcare costs.

Comparison: Patient outcomes, costs, and satisfaction will be evaluated, comparing patients assigned to follow-up using the Medtronic Carelink Monitor versus quarterly visits to an outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have an ICD with or without CRT for an approved indication
* Must be planning to have their devices followed-up at Duke
* Must have a telephone (land line)
* Willing and able to provide informed consent.

Exclusion Criteria:

* 18 years of age or younger
* No telephone with land line
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Re-hospitalization and ED visits for cardiac causes, unscheduled clinic visits for device-related issues, medications, patient logs, patients' level of satisfaction with their device care at baseline, 6 months, and 12 months. | 12 months

SECONDARY OUTCOMES:
Health-related quality of life at baseline, 6 months, and 12 months. Health utilization costs incurred during the study period. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sana Al-Khatib, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Al-Khatib SM, Piccini JP, Knight D, Stewart M, Clapp-Channing N, Sanders GD. Remote monitoring of implantable cardioverter defibrillators versus quarterly device interrogations in clinic: results from a randomized pilot clinical trial. J Cardiovasc Electrophysiol. 2010 May;21(5):545-50. doi: 10.1111/j.1540-8167.2009.01659.x. Epub 2009 Dec 15. PMID 20021522